CLINICAL TRIAL: NCT00700752
Title: A Comparison of Two Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0728
Record Dates: First submitted 2008-06-17; First posted 2008-06-19 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Refractive Error; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A/balafilcon A (Active Comparator): senofilcon A silicone hydrogel contact lens worn during first 4-week period, balafilcon A silicone hydrogel contact lens worn during the second 4-week period. Senofilcon A lenses worn daily on a 2-week replacement schedule; balafilcon A lenses worn daily on a 4-week replacement schedule. Lens replacement conducted in-office in a masked process.
  Interventions: Device: senofilcon A; Device: balafilcon A
- balafilcon A/senofilcon A (Active Comparator): balafilcon A silicone hydrogel contact lens worn worn during first 4-week period, senofilcon A silicone hydrogel contact lens worn during the second 4-week period. Senofilcon A lenses worn daily on a 2-week replacement schedule; balafilcon A lenses worn daily on a 4-week replacement schedule. Lens replacement conducted in-office in a masked process.
  Interventions: Device: senofilcon A; Device: balafilcon A

INTERVENTIONS:
Device: senofilcon A — silicone hydrogel contact lens
Device: balafilcon A — silicone hydrogel contact lens

SUMMARY:
This study seeks to evaluate the clinical and subjective performance of two established soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age (18 years) and capacity to volunteer.
2. They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They would be expected to attain at least 6/9 (20/30) in each eye with the study lenses.
5. They are able to wear contact lenses with a back vertex power of -1.00 to -6.00DS.
6. They have a maximum of 1.00D of refractive astigmatism (i.e. ≤ 1.00 DC).
7. They have successfully worn contact lenses within six months of starting the study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
7. They are pregnant or lactating.
8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
9. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV).
10. They have diabetes.
11. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Senofilcon A/Balafilcon A: senofilcon A silicone hydrogel contact lens worn first, balafilcon A silicone hydrogel contact lens worn second.
- Balafilcon A/Senofilcon A: balafilcon A silicone hydrogel contact lens worn first, senofilcon A silicone hydrogel contact lens worn second.
Period: First Intervention
Arm/Group | Senofilcon A/Balafilcon A | Balafilcon A/Senofilcon A
Started | 20 | 20
Completed | 20 | 18
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Intervention
Arm/Group | Senofilcon A/Balafilcon A | Balafilcon A/Senofilcon A
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Completed study population
Arm/Group | Overall
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Comfort at at the Manufacturer's Recommended Lens Replacement Timeframe of 2-weeks (Senofilcon A) or 4-weeks (Balafilcon A).
Description: Subjective rating of overall comfort using a 0 through 5 scale. 0=n/a, 1=poor, 2=fair, 3=good, 4=very good, 5=excellent. Scores from 2-week and 4-week visits were combined for final values.
Time Frame: after 4 weeks of lens wear
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Senofilcon A: silicone hydrogel contact lens worn daily with a 2-week replacement regimen.
- Balafilcon A: silicone hydrogel contact lens worn daily with a 4-week replacement regimen
Arm/Group | Senofilcon A | Balafilcon A
Number analyzed (Participants) | 38 | 38
Units on a scale | 4.0074 (0.2008) | 2.8438 (0.1972)
Statistical Analysis 1: Comparison: Senofilcon A vs Balafilcon A; Alternative hypothesis is senofilcon A is superior to balafilcon A for comfort; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.1636, 95% CI 2-sided [0.7890 to 1.1636], Standard Error of Mean 0.1887 — The mean difference is calculated as senofilcon A minus balafilcon A

ADVERSE EVENTS:
Arm/Group | Senofilcon A/Balafilcon A | Balafilcon A/Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.